CLINICAL TRIAL: NCT07345429
Title: ONE-YEAR OUTCOMES OF ANTHROPOMETRIC, BIOCHEMICAL, AND NUTRITIONAL PARAMETERS AFTER CONVERSION BARIATRIC SURGERY
Brief Title: One-Year Outcomes After Conversion Bariatric Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: Medipol University (Other)
Collaborators: Mudanya University (Other)
Responsible Party: Principal Investigator, Seher Şen, Assistant Professor, Principal Investigator, Mudanya University
Other Study IDs: MUDU-SBE-SS-01
Record Dates: First submitted 2025-12-17; First posted 2026-01-15 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Obesity & Overweight; Bariatric Surgery; Revisional Bariatric Surgery
Keywords: conversion bariatric surgery; obesity; nutritional assessment; weight regain; metabolic outcomes; anthropometric measurements
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Conversion Bariatric Surgery: This cohort includes patients who previously underwent conversion bariatric surgery as part of routine clinical care and were followed observationally. Anthropometric measurements, biochemical parameters, and nutritional status were assessed at the preoperative period and postoperative month 12 (1 year).

SUMMARY:
Obesity is a growing global public health problem, and bariatric surgery is currently the most effective treatment for achieving sustained weight loss and improving obesity-related comorbidities. However, a subset of patients experience inadequate weight loss or weight regain following primary bariatric surgery, which may lead to the recurrence of metabolic complications and reduced quality of life. In such cases, conversion bariatric surgery, defined as the surgical conversion from one bariatric procedure to another, is considered an important therapeutic option. Despite the increasing number of conversion procedures, comprehensive longitudinal data evaluating anthropometric, biochemical, and nutritional outcomes after conversion bariatric surgery remain limited.

This study aims to prospectively evaluate individuals undergoing conversion bariatric surgery due to weight regain following primary bariatric surgery. Anthropometric measurements, biochemical parameters, and nutritional status will be assessed preoperatively and at 1 year after surgery. By evaluating weight loss outcomes together with metabolic and nutritional changes, this study seeks to provide clinically relevant evidence to guide postoperative follow-up strategies, optimize nutritional management, and support multidisciplinary care in patients undergoing conversion bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-45 years
* Previously underwent bariatric surgery
* Subsequently underwent conversion bariatric surgery due to suboptimal clinical response

Suboptimal clinical response defined as either:

* Suboptimal Clinical Response (SCR): maximum total weight loss (TWL%) of <20% within 18 months after metabolic and bariatric surgery
* Recurrent Weight Gain (RWG): regaining >30% of initial postoperative weight loss after achieving initial weight reduction

Exclusion Criteria:

* Pregnancy or lactation
* Presence of acute illness or infection
* Comorbid conditions that could limit treatment efficacy or compromise safety
* Participation in professional athletic activity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18-65 years who had previously undergone bariatric surgery and subsequently received conversion bariatric surgery due to suboptimal clinical response, defined as suboptimal weight loss or recurrent weight gain. Participants are followed in routine clinical practice and evaluated preoperatively and at postoperative 1 year for anthropometric, biochemical, nutritional, and physical activity outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2026-01-10 (Actual); Study Completion 2026-02-21 (Estimated)

PRIMARY OUTCOMES:
Change in Body Composition Parameters | Preoperative baseline and postoperative 1 year
  Body composition parameters including fat mass, fat percentage, fat-free mass, fat-free mass percentage, skeletal muscle mass, muscle percentage, and extracellular water to total body water ratio assessed using multi-frequency bioelectrical impedance analysis (BIA).
Change in Body Weight | Preoperative baseline and postoperative 1 year
  Change in body weight (kg) measured using a digital scale with participants wearing light clothing and no shoes.
Change in Body Mass Index (BMI) | Preoperative baseline and postoperative 1 year
  Change in body mass index (kg/m²) calculated from measured body weight and height.
Percentage of Total Weight Loss | postoperative 1 year
  Percentage of total weight loss calculated as [(preoperative weight - postoperative weight) / preoperative weight] × 100.
Percentage of Excess Weight Loss | postoperative 1 year
  Percentage of excess weight loss calculated as [(preoperative weight - postoperative weight) / (preoperative weight - ideal body weight)] × 100, with ideal body weight defined as a BMI of 25 kg/m².
Change in Waist Circumference | Preoperative baseline and postoperative 1 year
  Waist circumference (cm) measured in the standing position using a non-elastic measuring tape at the midpoint between the lowest rib and the iliac crest.
Change in Hip Circumference | Preoperative baseline and postoperative 1 year
  Hip circumference (cm) measured in the standing position at the point of maximum protrusion of the gluteal muscles using a non-elastic measuring tape.
Change in Body Fat Percentage (%) | Preoperative baseline and postoperative 1 year
  Body fat percentage measured using multi-frequency bioelectrical impedance analysis (BIA).
Change in Fat-Free Mass (kg) | Preoperative baseline and postoperative 1 year
  Fat-free mass measured using multi-frequency bioelectrical impedance analysis (BIA).
Change in Skeletal Muscle Mass (kg) | Preoperative baseline and postoperative 1 year
  Skeletal muscle mass measured using multi-frequency bioelectrical impedance analysis (BIA).

SECONDARY OUTCOMES:
Change in Fasting Plasma Glucose | Preoperative baseline and postoperative 1 year
  Changes in fasting plasma glucose levels measured from venous blood samples.
Change in Alanine Aminotransferase (ALT) | Preoperative baseline and postoperative 1 year
  Changes in alanine aminotransferase (ALT) levels measured from venous blood samples.
Change in Hematological Parameters | Preoperative baseline and postoperative 1 year
  Changes in hemoglobin and hematocrit levels measured from venous blood samples.
Change in Iron Status Parameters | Preoperative baseline and postoperative 1 year
  Changes in serum ferritin, serum iron, and total iron-binding capacity levels measured from venous blood samples.
Change in Micronutrient and Electrolyte Levels | Preoperative baseline and postoperative 1 year
  Changes in serum vitamin B12, folic acid, magnesium, total calcium, sodium, and potassium levels measured from venous blood samples.
Change in Fasting Insulin | Preoperative baseline and postoperative 1 year
  Changes in fasting insulin levels measured from venous blood samples.
Change in Glycated Hemoglobin (HbA1c) | Preoperative baseline and postoperative 1 year
  Changes in glycated hemoglobin (HbA1c) levels measured from venous blood samples.
Change in Total Cholesterol | Preoperative baseline and postoperative 1 year
  Changes in total cholesterol levels measured from venous blood samples.
Change in LDL Cholesterol | Preoperative baseline and postoperative 1 year
  Changes in low-density lipoprotein (LDL) cholesterol levels measured from venous blood samples.
Change in HDL Cholesterol | Preoperative baseline and postoperative 1 year
  Changes in high-density lipoprotein (HDL) cholesterol levels measured from venous blood samples.
Change in Triglyceride Levels | Preoperative baseline and postoperative 1 year
  Changes in triglyceride levels measured from venous blood samples
Change in Aspartate Aminotransferase (AST) | Preoperative baseline and postoperative 1 year
  Changes in aspartate aminotransferase (AST) levels measured from venous blood samples.
Change in Urea Levels | Preoperative baseline and postoperative 1 year
  Changes in serum urea levels measured from venous blood samples.
Change in Uric Acid Levels | Preoperative baseline and postoperative 1 year
  Changes in serum uric acid levels measured from venous blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Seher Şen, Assistant Professor, Principal Investigator — Mudanya University
Locations (1):
- Mudanya Univesity, Osmangazi, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to the need to protect patient privacy and confidentiality.